CLINICAL TRIAL: NCT01683799
Title: Slow Wave Sleep and Inflammatory Processes in Pain
Brief Title: Sleep, Pain and Inflammatory Processes in Older Adults With Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kathi Heffner, Associate Professor of Psychiatry, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RSRB00044088; R21AG041942-01A1 (NIH)
Record Dates: First submitted 2012-09-07; First posted 2012-09-12 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Osteoarthritis of the Knee; Insomnia; Knee Pain
Keywords: Osteoarthritis; Insomnia; Chronic pain; Cognitive Behavioral Therapy for Insomnia; Inflammation; Inflammatory cytokines
MeSH Terms: conditions — Osteoarthritis, Knee; Sleep Initiation and Maintenance Disorders; Osteoarthritis; Chronic Pain; Inflammation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insomnia treatment (Experimental): Cognitive Behavioral Therapy for Insomnia
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — 6-week behavioral treatment for insomnia
  Arms: Insomnia treatment

SUMMARY:
The purpose if the study is to determine whether improving sleep, especially slow wave or "deep" sleep, in older adults with osteoarthritis (OA) and insomnia reduces pain sensitivity and inflammatory responses to pain, and improves OA-related pain.

ELIGIBILITY:
Inclusion Criteria:

* 50-75 years of age (for women, post-menopausal)
* Kellgren-Lawrence grade II radiographic evidence of OA affecting one or both knees
* knee pain on most days for ≥ 6 months
* self-reported disability due to knee pain for ≥ 2 of the following: walking, kneeling, ascending or descending stairs, or performing daily activities
* willing and able to avoid all prescription and non-prescription, non-opiate pain medication for 48 hours prior to testing and all narcotic pain medication for 2 weeks prior to testing
* meets research diagnostic criteria for sleep maintenance insomnia

Exclusion Criteria:

* health conditions with immunological components or undergoing or taking immunosuppressive therapies
* conditions contraindicated for or potentially limiting ability to conduct NFR and/or cold pressor test (e.g. Raynaud's syndrome; seizures; prior MI; respiratory conditions; leg/hip nerve damage; BMI ≥ 32)
* sleep disorders other than insomnia
* dementia or cognitive impairment
* history of schizophrenia or bipolar I disorder; current or recent history (within 3 months) of major psychiatric disorders
* current depressive symptomatology or current suicidality
* active substance dependence
* untreated hypertension
* use of antidepressants (stable use for 3 months okay), antipsychotics, mood stabilizers, sedative-hypnotics, opiate analgesics

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-02; Primary Completion 2015-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in minutes of time in slow wave sleep | baseline and 10 weeks
Change from baseline in relative power of delta EEG activity to index slow wave sleep activity | baseline and 10 weeks
Change from baseline in nociception flexion reflex threshold | baseline and 10 weeks
Change from baseline in electrocutaneous pain threshold | baseline and 10 weeks
Change from baseline in inflammatory cytokine responses to pain | baseline and 10 weeks
Change from baseline in Western Ontario and McMaster University OA Index | baseline and 10 weeks
Change from baseline in Knee Pain Scale score | baseline and 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathi L. Heffner, PhD, Principal Investigator — University of Rochester; Wilfred Pigeon, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States